CLINICAL TRIAL: NCT05865002
Title: A Phase 1, Open Label, Dose Escalation, Dose Expansion, Multicenter, First in Human Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics of Oral AUR107 in Patients With Relapsed Advanced Malignancies (SHAKTI-1)
Brief Title: A Study Evaluating the Safety and Efficacy of AUR107 in Patients With Relapsed Advanced Malignancies (SHAKTI-1)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aurigene Discovery Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AUR107-101
Record Dates: First submitted 2023-04-28; First posted 2023-05-18 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-05

CONDITIONS: Relapsed Malignant Solid Neoplasm
Keywords: Relapse malignant neoplasm; Non small cell lung cancer; Gastric cancer; Colon cancer; Esophageal cancer; Kidney cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Colonic Neoplasms; Esophageal Neoplasms; Kidney Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose Escalation "3+3" Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AUR107, 5mg to 200mg (Experimental): Currently, planned dose levels are 5 mg QD, 10 mg QD, 20 mg QD, 40 mg QD, 60 mg QD, 90 mg QD, 135 mg QD, and 200 mg QD
  Interventions: Drug: AUR107

INTERVENTIONS:
Drug: AUR107 — Once daily

SUMMARY:
An open-label, first-in-human, Phase 1 study in adult patients with relapsed advanced malignancies will be done to assess AUR107 safety, tolerability, pharmacokinetics, pharmacodynamics, and optimal biological dose.

DETAILED DESCRIPTION:
This is a Phase I, Open Label, Dose-Escalation, First-in-Human study in adult patients with select relapsed advanced malignancies. The safety and tolerability of oral AUR107 will be evaluated in patients with selected advanced solid tumors (Non-small cell lung cancer, Gastric cancer, Urothelial cancer, Kidney cancer, Colon cancer, and Esophageal cancer) who do not have any available curative or life-prolonging treatment options and have exhausted all effective locally available therapies. The traditional 3+3 design for dose escalation will be used to evaluate the safety, pharmacokinetics/pharmacodynamics, and determine the Optimal Biological Dose of AUR107 as a single agent. The Optimal Biological Dose will be selected using a totality of safety, PK, and PD data.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years of age.
2. Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1.
3. Acceptable bone marrow and organ function at screening as described below:

   1. ANC ≥ 1500/μL (without WBC growth factor support)
   2. Platelet count ≥ 100,000/μL without transfusion support
   3. Hemoglobin ≥ 9 g/dL (Transfusion is allowed to achieve this Hb)
   4. Total Bilirubin ≤ 1.5 x ULN; (Patients with known Gilbert's syndrome are allowed with a Total Bilirubin ≤ 2.5 x ULN)
   5. AST (SGOT) ≤ 3 x ULN (≤ 5 × ULN if known liver metastases)
   6. ALT (SGPT) ≤ 3 x ULN (≤ 5 × ULN if known liver metastases)
   7. Creatinine clearance (CrCl) ≥ 60 mL/min (either measured or estimated by the Cockcroft-Gault formula).
4. Ability to swallow and retain oral medications.
5. Histopathological diagnosis of a solid tumor. Note: The solid tumors must be in Stage IV at screening.
6. Evidence of measurable disease per RECIST, v1.1 for solid tumors.
7. Standard curative measures do not exist, and the patient must have exhausted all effective therapies available locally.

Notes:

7a. At a minimum, solid tumor patients must have received at least two lines of systemic therapies in the metastatic incurable settings (these two lines must be in the metastatic setting and not in the earlier stage of cancer).

7b. Any cancer patient with access to any effective therapy must not be enrolled

Exclusion Criteria:

1. Systemic anti-cancer therapy, such as chemotherapy, biological therapy, or immunomodulatory drug therapy, received within the past 28 days or 5 half-lives, whichever is longer, from Cycle 1 Day 1 of the study.

   Note: Concomitant use of low-dose prednisone (up to 10 mg/day) or medroxyprogesterone is allowed.

   Note: Patients with CRPC (castrate-resistant prostate cancer) should continue to receive ongoing medical castration with LHRH analogs, and such patients are allowed.
2. Presence of acute or chronic toxicity resulting from prior anticancer treatment, with the exception of alopecia or nail changes, that has not resolved to Grade ≤ 1, as determined by NCI CTCAE v 5.0.
3. Definitive Radiotherapy within the last 21 days of Cycle 1 Day 1 (limited field palliative radiation is allowed and no restrictions during the screening period or during the trial)

   • Use of any investigational agent within 28 days or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1.
4. Use of drugs which are moderate / strong CYP3A4 inducers and/or drugs which are predominantly metabolized by CYP3A4 within 1week or 5 half-lives (whichever is longer) prior to Cycle 1 Day 1.

   • Note: This class of drugs are also prohibited during DLT evaluation period and must be either avoided or used with caution beyond DLT evaluation period.
5. Known symptomatic or untreated or recently treated (≤ 6 months of screening) central nervous system (CNS) metastases. Patients with previously treated (> 6 months of screening) CNS metastases and are now stable and asymptomatic, from CNS perspective, are allowed.
6. Major surgery ≤ 28 days from Cycle 1 Day 1 (major surgery is defined as a procedure requiring general anesthesia).
7. Patients with leukemia, myelodysplastic syndrome, multiple myeloma, or lymphoma.
8. Active infection requiring systemic therapy. Note: Prophylactic use of antibiotics is allowed. Any infection detected during the screening period which is resolved adequately according to investigator before the Cycle 1 Day 1, is allowed.
9. Known to be human immunodeficiency virus (HIV) positive or have an acquired immunodeficiency syndrome-related illness.
10. Known active or chronic hepatitis B (HBsAg +ve) or hepatitis C infection (HCV antibody +ve).
11. The patient who is expected to require any other form of antineoplastic therapy or targeted therapy while on study.
12. Uncontrolled congestive heart failure (New York Heart Association [NYHA] Class 2-4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, or transient ischemic attack, or pulmonary embolism within 3 months prior to Cycle 1 Day 1.
13. Ongoing cardiac dysrhythmias requiring treatment of any grade or treatment of cardiac dysrhythmias in the past 3 months, before Cycle 1 Day 1.
14. QTc (Bazzett) interval >460 ms on ECG at screening and/or at Cycle 1 Day 1 pre-dose.
15. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or significant gastritis, active bleeding diatheses, presence of any major medical illness (e.g., renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, or psychiatric illness/social situations or clinically significant laboratory / ECG abnormalities at screening, any or a combination of illnesses, which, in the opinion of the PI, may either put the patient at risk because of participation in the study or influence the results or the patient's ability to participate in the study.
16. Current swab-positive or suspected (under investigation) Covid-19 infection or fever and other signs or symptoms suggestive of Covid-19 infection with recent contact of the person(s) with confirmed Covid-19 infection, at screening or Day 1 of Cycle 1.
17. Positive pregnancy test for women of childbearing potential (WOCBP) at the screening or enrolment visit.
18. Lactating women or WOCBP who are neither surgically sterilized nor willing to use reliable contraceptive methods. (hormonal contraceptive, IUD, or any double combination of the male or female condom, spermicidal gel, diaphragm, sponge, cervical cap).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
First cycle Dose Limiting Toxicities (DLT) | 28 days
  Assess dose limiliting toxicities of AUR107
Safety of AUR107 as measured by the number of participants with treatment-related adverse events (AE) graded according to NCI CTCAE version 5.0 | 28 days
  The assessment of safety was based on the frequency of deaths, AEs, SAEs, AEs leading to discontinuation of study drug, and abnormalities in specific clinical laboratory assessments. AEs and laboratory values will be graded for severity according to the NCI CTCAE version 5.0.
Optimal Biological Dose | 28 days
  Determine optimal Biological dose
Pharmacokinetics: Maximum concentration (Cmax) | Day 1 and Day 15
  Maximum concentration of AUR107
Pharmacokinetics: Time to Maximum concentration (Tmax) | Day 1 and Day 15
  Tmax in hours
Pharmacokinetics: Area under the curve (AUC) | Day 1 and Day 15
  Area under the curve (AUC) of AUR 107 in h* mcg/mL
Pharmacokinetics: Mean Residence Time (MRT) | Day 1 and Day 15
  Average time the drugs stays in the body
Pharmacokinetics: Terminal elimination half-life | Day 1 and Day 15
  Terminal elimination half-life of AUR 107 in hours
Maximum concentration (Cmax) administered under fasting/fed condition | Day 8 and Day 9
  Compare in fast and fed conditions
Time to Maximum concentration (Tmax) administered under fasting/fed condition | Day 8 and Day 9
  Compare Tmax in fast and fed conditions
Area under curve (AUC) administered under fasting/fed condition | Day 8 and Day 9
  Compare AUC in fast and fed conditions

OTHER OUTCOMES:
Exploratory endpoint: Identification of gene expression profiles | Day 1, Day 2, and Day 15
  Pharmacodynamic marker: Gene Expression profile as assessed by RNA analysis
Exploratory endpoint- Efficacy assessments, Overall Response Rate | Through study completion, an average of 1 year
  Efficacy assessments-Overall Response Rate
Exploratory endpoint- Efficacy assessments, Duration of Response | Through study completion, an average of 1 year
  Efficacy assessments- Duration of Response
Exploratory endpoint- Efficacy assessments, Progression Free Survival (PFS) | Through study completion, an average of 1 year
  Efficacy assessments- Progression Free Survival (PFS)
Median Change from Baseline to End of Treatment in Tumor-Specific Markers, CA-125 in ovarian cancer | Through study completion, an average of 1 year
  Change in Tumor Specific Markers - CA-125 in ovarian cancer
Median Change from Baseline to End of Treatment in Tumor-Specific Markers, PSA in Castrate Resistant Prostate Cancer | Through study completion, an average of 1 year
  Change in Tumor Specific Markers - PSA in Castrate Resistant Prostate Cancer
Median Change from Baseline to End of Treatment in Tumor-Specific Markers, CEA in colorectal cancer | Through study completion, an average of 1 year
  Change in Tumor Specific Markers - CEA in colorectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Akhil Kumar, Principal Investigator — Aurigene Oncology Limited
Locations (8):
- India (8):
  - HCG City Cancer Centre, Vijayawada, Andhra Pradesh
  - Omega Hospital, Visakhapatnam, Andhra Pradesh
  - Unique Hospital Multispeciality and Research Institute, Surat, Gujarat
  - Vydehi Institute of Medical Sciences and Research Centre, Bangalore, Karnataka
  - K R Hospital, Mysore, Karnataka
  - Krupamayi Hospital, Aurangabad, Maharashtra
  - Grant Medical Foundation Ruby Hall Clinic, Pune, Maharashtra
  - All India Institute of Medical Sciences, New Delhi

IPD SHARING:
Plan to Share IPD: No